CLINICAL TRIAL: NCT07002294
Title: The Effect of SPecialty cAre on Recovery From Cardiac Arrest Trial (the SPARC Trial)
Acronym: SPARC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jonathan Elmer, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25050152; R61HL175113 (NIH)
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest (CA); Heart Arrest; Heart Arrest, Out-Of-Hospital
Keywords: cardiac arrest
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transfer to specialty care (Experimental): Participants randomized to receive specialty care will undergo immediate interfacility transport to and hospital treatment at the specialty care hospital
  Interventions: Other: Transfer to specialty care
- Usual care (Active Comparator): Participants randomized to the usual care arm will be hospitalized at the first hospital or transferred to the closest appropriate hospital
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Transfer to specialty care — Interfacility transport and treatment at the specialty care hospital
  Arms: Transfer to specialty care
Other: Usual care — Hospitalization and treatment at the closest appropriate facility
  Arms: Usual care

SUMMARY:
This randomized clinical trial will determine if adult participants who are in the emergency department after being resuscitated from a cardiac arrest outside of the hospital benefit from care delivered at specialized centers.

The main question that it will answer is whether transferring participants to a hospital with a specialized cardiac arrest service improves recovery of function after 90 days.

Participants will receive all usual medical care, but some participants will be offered transfer to a regional cardiac arrest center and others will be offered care at the closest appropriate hospital. Investigators will interview participants after 90 days to assess their recovery.

DETAILED DESCRIPTION:
Cardiac arrest is a sudden stopping of the heart, which can sometimes be reversed by rapid cardiopulmonary resuscitation (CPR) and emergency medical care. Each year, over 150,000 Americans are admitted to the hospital after receiving CPR. However, many of these patients die in the hospital. There is wide variation in patient outcomes between hospitals. A key knowledge gap about systems of care is whether specific hospital or subsequent interventions or processes of care are associated with better patient outcomes. Specifically, it is unknown if patient outcomes are improved by specialized centers or by improved implementation of recommended interventions at all hospitals.

Observational data in our region and internationally suggest that out-of-hospital cardiac arrest outcomes are better when patients who survive CPR are hospitalized in specialty care or high-volume centers. It is unclear from these studies what are the minimal capabilities that distinguish specialty care from usual care and which aspects of specialty care are influencing outcomes.

This trial will take advantage of a regional system of care that includes 18 hospitals in southwestern Pennsylvania that treat over 1,000 patients resuscitated from out-of-hospital cardiac arrest annually. This region includes one high-volume specialty center with specific attention to recommended interventions for this patient population, as well as several secondary and tertiary care facilities with variable resources and approaches to patient care. This randomized trial will compare outcomes for patients assigned to care at the specialty center versus other centers and will leverage the heterogeneity of treatment between centers to understand the influence of specific treatments.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest
* Resuscitated from cardiac arrest with palpable pulse in the emergency department
* Treated at one of participating hospital emergency departments
* Age ≥18 years

Exclusion Criteria:

* Known prior advanced directives or decision to limit critical care
* Known pre-arrest dependent functional status (e.g., living in a skilled nursing facility, hospice or bedbound)
* Arrest in the emergency department >4 hours after arrival
* Traumatic etiology of arrest
* Known to have opted-out from the SPARC trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1618 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2031-06 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | 90 Days post arrest
  The Modified Rankin Scale (mRS) is a measure of functional recovery, measured 90 days after cardiac arrest. A Modified Rankin Score (mRS) of 0 corresponds to full functional recovery and a Modified Rankin Score (mRS) of 6 corresponds to death, with progressively worse functional outcomes at higher scores. Intermediate values reflect progressive functional dependence, with higher scores reflecting greater dependence on others.

SECONDARY OUTCOMES:
Survival to ICU Admission | 24 hours post arrest
72 hour survival | 72 hours post arrest
mRS at hospital discharge | Up to 6 months post arrest

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Elmer, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Department of Emergency Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data may be shared in the future with investigators at other institutions. The local investigators will execute data use agreements with outside investigators and institutions prior to sharing any data. Identifiable data will not be shared.

REFERENCES:
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Elmer J, Weisgerber AR, Wallace DJ, Horne E, Stuart SA, Shutterly K, Callaway CW. Between-hospital variability in organ donation after resuscitation from out-of-hospital cardiac arrest. Resuscitation. 2021 Oct;167:372-379. doi: 10.1016/j.resuscitation.2021.07.038. Epub 2021 Aug 4. PMID 34363855
- [Background] Elmer J, Molyneaux BJ, Shutterly K, Stuart SA, Callaway CW, Darby JM, Weisgerber AR. Organ donation after resuscitation from cardiac arrest. Resuscitation. 2019 Dec;145:63-69. doi: 10.1016/j.resuscitation.2019.10.013. Epub 2019 Oct 22. PMID 31654724
- [Background] Imai K, Keele L, Tingley D. A general approach to causal mediation analysis. Psychol Methods. 2010 Dec;15(4):309-34. doi: 10.1037/a0020761. PMID 20954780
- [Background] VanderWeele TJ. A unification of mediation and interaction: a 4-way decomposition. Epidemiology. 2014 Sep;25(5):749-61. doi: 10.1097/EDE.0000000000000121. PMID 25000145
- [Background] VanderWeele TJ. Bias formulas for sensitivity analysis for direct and indirect effects. Epidemiology. 2010 Jul;21(4):540-51. doi: 10.1097/EDE.0b013e3181df191c. PMID 20479643
- [Background] VanderWeele TJ. Commentary: On Causes, Causal Inference, and Potential Outcomes. Int J Epidemiol. 2016 Dec 1;45(6):1809-1816. doi: 10.1093/ije/dyw230. No abstract available. PMID 28130319
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Kahan BC, Jairath V, Dore CJ, Morris TP. The risks and rewards of covariate adjustment in randomized trials: an assessment of 12 outcomes from 8 studies. Trials. 2014 Apr 23;15:139. doi: 10.1186/1745-6215-15-139. PMID 24755011
- [Background] Elmer J, Coppler PJ, May TL, Hirsch K, Faro J, Solanki P, Brown M, Puyana JS, Rittenberger JC, Callaway CW. Unsupervised learning of early post-arrest brain injury phenotypes. Resuscitation. 2020 Aug;153:154-160. doi: 10.1016/j.resuscitation.2020.05.051. Epub 2020 Jun 9. PMID 32531403
- [Background] Callaway CW, Schmicker R, Kampmeyer M, Powell J, Rea TD, Daya MR, Aufderheide TP, Davis DP, Rittenberger JC, Idris AH, Nichol G; Resuscitation Outcomes Consortium (ROC) Investigators. Receiving hospital characteristics associated with survival after out-of-hospital cardiac arrest. Resuscitation. 2010 May;81(5):524-9. doi: 10.1016/j.resuscitation.2009.12.006. Epub 2010 Jan 13. PMID 20071070
- [Background] Campbell BCV, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Dowling RJ, Yan B, Bush SJ, Dewey HM, Thijs V, Scroop R, Simpson M, Brooks M, Asadi H, Wu TY, Shah DG, Wijeratne T, Ang T, Miteff F, Levi CR, Rodrigues E, Zhao H, Salvaris P, Garcia-Esperon C, Bailey P, Rice H, de Villiers L, Brown H, Redmond K, Leggett D, Fink JN, Collecutt W, Wong AA, Muller C, Coulthard A, Mitchell K, Clouston J, Mahady K, Field D, Ma H, Phan TG, Chong W, Chandra RV, Slater LA, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Bladin CF, Sharma G, Desmond PM, Parsons MW, Donnan GA, Davis SM; EXTEND-IA TNK Investigators. Tenecteplase versus Alteplase before Thrombectomy for Ischemic Stroke. N Engl J Med. 2018 Apr 26;378(17):1573-1582. doi: 10.1056/NEJMoa1716405. PMID 29694815
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Background] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Background] Peterson B, Harrell FE. Partial Proportional Odds Models for Ordinal Response Variables. Journal of the Royal Statistical Society Series C (Applied Statistics) 1990;39:205-17
- [Background] Janssen PM, Visser NA, Dorhout Mees SM, Klijn CJ, Algra A, Rinkel GJ. Comparison of telephone and face-to-face assessment of the modified Rankin Scale. Cerebrovasc Dis. 2010 Jan;29(2):137-9. doi: 10.1159/000262309. Epub 2009 Dec 1. PMID 19955737
- [Background] Haywood K, Whitehead L, Nadkarni VM, Achana F, Beesems S, Bottiger BW, Brooks A, Castren M, Ong ME, Hazinski MF, Koster RW, Lilja G, Long J, Monsieurs KG, Morley PT, Morrison L, Nichol G, Oriolo V, Saposnik G, Smyth M, Spearpoint K, Williams B, Perkins GD; COSCA Collaborators. COSCA (Core Outcome Set for Cardiac Arrest) in Adults: An Advisory Statement From the International Liaison Committee on Resuscitation. Circulation. 2018 May 29;137(22):e783-e801. doi: 10.1161/CIR.0000000000000562. Epub 2018 Apr 26. PMID 29700122
- [Background] Zadorozny EV, Guyette FX, Flickinger KL, Martin-Gill C, Amoah K, Artist O, Mohammed A, Condle JP, Callaway CW, Elmer J, Coppler PJ; Pittsburgh Post Cardiac Arrest Service. Time to specialty care and mortality after cardiac arrest. Am J Emerg Med. 2021 Dec;50:618-624. doi: 10.1016/j.ajem.2021.09.044. Epub 2021 Sep 23. PMID 34879476
- [Background] Morrison LJ, Nichol G, Rea TD, Christenson J, Callaway CW, Stephens S, Pirrallo RG, Atkins DL, Davis DP, Idris AH, Newgard C; ROC Investigators. Rationale, development and implementation of the Resuscitation Outcomes Consortium Epistry-Cardiac Arrest. Resuscitation. 2008 Aug;78(2):161-9. doi: 10.1016/j.resuscitation.2008.02.020. Epub 2008 May 13. PMID 18479802
- [Background] Elmer J, Callaway CW, Chang CH, Madaras J, Martin-Gill C, Nawrocki P, Seaman KAC, Sequeira D, Traynor OT, Venkat A, Walker H, Wallace DJ, Guyette FX. Long-Term Outcomes of Out-of-Hospital Cardiac Arrest Care at Regionalized Centers. Ann Emerg Med. 2019 Jan;73(1):29-39. doi: 10.1016/j.annemergmed.2018.05.018. Epub 2018 Jul 4. PMID 30060961
- [Background] Elmer J, Gianakas JJ, Rittenberger JC, Baldwin ME, Faro J, Plummer C, Shutter LA, Wassel CL, Callaway CW, Fabio A; Pittsburgh Post-Cardiac Arrest Service. Group-Based Trajectory Modeling of Suppression Ratio After Cardiac Arrest. Neurocrit Care. 2016 Dec;25(3):415-423. doi: 10.1007/s12028-016-0263-9. PMID 27033709
- [Background] Rittenberger JC, Guyette FX, Tisherman SA, DeVita MA, Alvarez RJ, Callaway CW. Outcomes of a hospital-wide plan to improve care of comatose survivors of cardiac arrest. Resuscitation. 2008 Nov;79(2):198-204. doi: 10.1016/j.resuscitation.2008.08.014. PMID 18951113
- [Background] Perkins GD, Jacobs IG, Nadkarni VM, Berg RA, Bhanji F, Biarent D, Bossaert LL, Brett SJ, Chamberlain D, de Caen AR, Deakin CD, Finn JC, Grasner JT, Hazinski MF, Iwami T, Koster RW, Lim SH, Huei-Ming Ma M, McNally BF, Morley PT, Morrison LJ, Monsieurs KG, Montgomery W, Nichol G, Okada K, Eng Hock Ong M, Travers AH, Nolan JP; Utstein Collaborators. Cardiac arrest and cardiopulmonary resuscitation outcome reports: update of the Utstein Resuscitation Registry Templates for Out-of-Hospital Cardiac Arrest: a statement for healthcare professionals from a task force of the International Liaison Committee on Resuscitation (American Heart Association, European Resuscitation Council, Australian and New Zealand Council on Resuscitation, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Southern Africa, Resuscitation Council of Asia); and the American Heart Association Emergency Cardiovascular Care Committee and the Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation. Circulation. 2015 Sep 29;132(13):1286-300. doi: 10.1161/CIR.0000000000000144. Epub 2014 Nov 11. PMID 25391522
- [Background] Elmer J, Dougherty M, Guyette FX, Martin-Gill C, Drake CD, Callaway CW, Wallace DJ. Comparing strategies for prehospital transport to specialty care after cardiac arrest. Resuscitation. 2023 Oct;191:109943. doi: 10.1016/j.resuscitation.2023.109943. Epub 2023 Aug 23. PMID 37625579
- [Background] Flickinger KL, Jaramillo S, Repine MJ, Koller AC, Holm M, Skidmore E, Callaway C, Rittenberger JC. One-year outcomes in individual domains of the cerebral performance category extended. Resusc Plus. 2021 Dec 6;8:100184. doi: 10.1016/j.resplu.2021.100184. eCollection 2021 Dec. PMID 34934994
- [Background] Sawyer KN, Camp-Rogers TR, Kotini-Shah P, Del Rios M, Gossip MR, Moitra VK, Haywood KL, Dougherty CM, Lubitz SA, Rabinstein AA, Rittenberger JC, Callaway CW, Abella BS, Geocadin RG, Kurz MC; American Heart Association Emergency Cardiovascular Care Committee; Council on Cardiovascular and Stroke Nursing; Council on Genomic and Precision Medicine; Council on Quality of Care and Outcomes Research; and Stroke Council. Sudden Cardiac Arrest Survivorship: A Scientific Statement From the American Heart Association. Circulation. 2020 Mar 24;141(12):e654-e685. doi: 10.1161/CIR.0000000000000747. Epub 2020 Feb 12. PMID 32078390
- [Background] Sawyer KN, Callaway CW, Wagner AK. Life After Death: Surviving Cardiac Arrest-an Overview of Epidemiology, Best Acute Care Practices, and Considerations for Rehabilitation Care. Current Physical Medicine and Rehabilitation Reports 2017;5:30-9
- [Background] May TL, Ruthazer R, Riker RR, Friberg H, Patel N, Soreide E, Hand R, Stammet P, Dupont A, Hirsch KG, Agarwal S, Wanscher MJ, Dankiewicz J, Nielsen N, Seder DB, Kent DM. Early withdrawal of life support after resuscitation from cardiac arrest is common and may result in additional deaths. Resuscitation. 2019 Jun;139:308-313. doi: 10.1016/j.resuscitation.2019.02.031. Epub 2019 Mar 2. PMID 30836171
- [Background] Elmer J, Torres C, Aufderheide TP, Austin MA, Callaway CW, Golan E, Herren H, Jasti J, Kudenchuk PJ, Scales DC, Stub D, Richardson DK, Zive DM; Resuscitation Outcomes Consortium. Association of early withdrawal of life-sustaining therapy for perceived neurological prognosis with mortality after cardiac arrest. Resuscitation. 2016 May;102:127-35. doi: 10.1016/j.resuscitation.2016.01.016. Epub 2016 Feb 3. PMID 26836944
- [Background] Steinberg A, Grayek E, Arnold RM, Callaway C, Fischhoff B, Krishnamurti T, Mohan D, White DB, Elmer J. Physicians' cognitive approach to prognostication after cardiac arrest. Resuscitation. 2022 Apr;173:112-121. doi: 10.1016/j.resuscitation.2022.01.001. Epub 2022 Jan 8. PMID 35017011
- [Background] Moseby-Knappe M, Westhall E, Backman S, Mattsson-Carlgren N, Dragancea I, Lybeck A, Friberg H, Stammet P, Lilja G, Horn J, Kjaergaard J, Rylander C, Hassager C, Ullen S, Nielsen N, Cronberg T. Performance of a guideline-recommended algorithm for prognostication of poor neurological outcome after cardiac arrest. Intensive Care Med. 2020 Oct;46(10):1852-1862. doi: 10.1007/s00134-020-06080-9. Epub 2020 Jun 3. PMID 32494928
- [Background] Elmer J, Steinberg A, Callaway CW. Paucity of neuroprognostic testing after cardiac arrest in the United States. Resuscitation. 2023 Jul;188:109762. doi: 10.1016/j.resuscitation.2023.109762. Epub 2023 Mar 15. PMID 36924822
- [Background] Suen CG, Wood AJ, Burke JF, Betjemann JP, Guterman EL. Hospital EEG Capability and Associations With Interhospital Transfer in Status Epilepticus. Neurol Clin Pract. 2023 Apr;13(2):e200143. doi: 10.1212/CPJ.0000000000200143. Epub 2023 Mar 16. PMID 37064585
- [Background] Callaway CW, Donnino MW, Fink EL, Geocadin RG, Golan E, Kern KB, Leary M, Meurer WJ, Peberdy MA, Thompson TM, Zimmerman JL. Part 8: Post-Cardiac Arrest Care: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S465-82. doi: 10.1161/CIR.0000000000000262. No abstract available. PMID 26472996
- [Background] Duncan PW, Bushnell C, Sissine M, Coleman S, Lutz BJ, Johnson AM, Radman M, Pvru Bettger J, Zorowitz RD, Stein J. Comprehensive Stroke Care and Outcomes: Time for a Paradigm Shift. Stroke. 2021 Jan;52(1):385-393. doi: 10.1161/STROKEAHA.120.029678. Epub 2020 Dec 22. PMID 33349012
- [Background] Uffen JW, Oosterheert JJ, Schweitzer VA, Thursky K, Kaasjager HAH, Ekkelenkamp MB. Interventions for rapid recognition and treatment of sepsis in the emergency department: a narrative review. Clin Microbiol Infect. 2021 Feb;27(2):192-203. doi: 10.1016/j.cmi.2020.02.022. Epub 2020 Feb 29. PMID 32120030
- [Background] Sebat F, Musthafa AA, Johnson D, Kramer AA, Shoffner D, Eliason M, Henry K, Spurlock B. Effect of a rapid response system for patients in shock on time to treatment and mortality during 5 years. Crit Care Med. 2007 Nov;35(11):2568-75. doi: 10.1097/01.CCM.0000287593.54658.89. PMID 17901831
- [Background] Solanki P, Coppler PJ, Kvaloy JT, Baldwin MA, Callaway CW, Elmer J; Pittsburgh Post-Cardiac Arrest Service. Association of antiepileptic drugs with resolution of epileptiform activity after cardiac arrest. Resuscitation. 2019 Sep;142:82-90. doi: 10.1016/j.resuscitation.2019.07.007. Epub 2019 Jul 17. PMID 31325554
- [Background] Elmer J, Coppler PJ, Solanki P, Westover MB, Struck AF, Baldwin ME, Kurz MC, Callaway CW. Sensitivity of Continuous Electroencephalography to Detect Ictal Activity After Cardiac Arrest. JAMA Netw Open. 2020 Apr 1;3(4):e203751. doi: 10.1001/jamanetworkopen.2020.3751. PMID 32343353
- [Background] Nishikimi M, Ogura T, Nishida K, Hayashida K, Emoto R, Matsui S, Matsuda N, Iwami T. Outcome Related to Level of Targeted Temperature Management in Postcardiac Arrest Syndrome of Low, Moderate, and High Severities: A Nationwide Multicenter Prospective Registry. Crit Care Med. 2021 Aug 1;49(8):e741-e750. doi: 10.1097/CCM.0000000000005025. PMID 33826582
- [Background] Callaway CW, Coppler PJ, Faro J, Puyana JS, Solanki P, Dezfulian C, Doshi AA, Elmer J, Frisch A, Guyette FX, Okubo M, Rittenberger JC, Weissman A. Association of Initial Illness Severity and Outcomes After Cardiac Arrest With Targeted Temperature Management at 36 degrees C or 33 degrees C. JAMA Netw Open. 2020 Jul 1;3(7):e208215. doi: 10.1001/jamanetworkopen.2020.8215. PMID 32701158
- [Background] Perman SM, Bartos JA, Del Rios M, Donnino MW, Hirsch KG, Jentzer JC, Kudenchuk PJ, Kurz MC, Maciel CB, Menon V, Panchal AR, Rittenberger JC, Berg KM; American Heart Association Emergency Cardiovascular Care Committee, Council on Cardiovascular Surgery and Anesthesia; Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Peripheral Vascular Disease; Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation, and Stroke Council. Temperature Management for Comatose Adult Survivors of Cardiac Arrest: A Science Advisory From the American Heart Association. Circulation. 2023 Sep 19;148(12):982-988. doi: 10.1161/CIR.0000000000001164. Epub 2023 Aug 16. PMID 37584195
- [Background] Chen N, Callaway CW, Guyette FX, Rittenberger JC, Doshi AA, Dezfulian C, Elmer J; Pittsburgh Post-Cardiac Arrest Service. Arrest etiology among patients resuscitated from cardiac arrest. Resuscitation. 2018 Sep;130:33-40. doi: 10.1016/j.resuscitation.2018.06.024. Epub 2018 Jun 22. PMID 29940296
- [Background] Trzeciak S, Jones AE, Kilgannon JH, Milcarek B, Hunter K, Shapiro NI, Hollenberg SM, Dellinger P, Parrillo JE. Significance of arterial hypotension after resuscitation from cardiac arrest. Crit Care Med. 2009 Nov;37(11):2895-903; quiz 2904. doi: 10.1097/ccm.0b013e3181b01d8c. PMID 19866506
- [Background] Hartke A, Mumma BE, Rittenberger JC, Callaway CW, Guyette FX. Incidence of re-arrest and critical events during prolonged transport of post-cardiac arrest patients. Resuscitation. 2010 Aug;81(8):938-42. doi: 10.1016/j.resuscitation.2010.04.012. Epub 2010 May 21. PMID 20483520
- [Background] Elmer J, Scutella M, Pullalarevu R, Wang B, Vaghasia N, Trzeciak S, Rosario-Rivera BL, Guyette FX, Rittenberger JC, Dezfulian C; Pittsburgh Post-Cardiac Arrest Service (PCAS). The association between hyperoxia and patient outcomes after cardiac arrest: analysis of a high-resolution database. Intensive Care Med. 2015 Jan;41(1):49-57. doi: 10.1007/s00134-014-3555-6. Epub 2014 Dec 4. PMID 25472570
- [Background] Wang HE, Prince DK, Drennan IR, Grunau B, Carlbom DJ, Johnson N, Hansen M, Elmer J, Christenson J, Kudenchuk P, Aufderheide T, Weisfeldt M, Idris A, Trzeciak S, Kurz M, Rittenberger JC, Griffiths D, Jasti J, May S; Resuscitation Outcomes Consortium (ROC) Investigators. Post-resuscitation arterial oxygen and carbon dioxide and outcomes after out-of-hospital cardiac arrest. Resuscitation. 2017 Nov;120:113-118. doi: 10.1016/j.resuscitation.2017.08.244. Epub 2017 Sep 21. PMID 28870720
- [Background] Salcido DD, Stephenson AM, Condle JP, Callaway CW, Menegazzi JJ. Incidence of rearrest after return of spontaneous circulation in out-of-hospital cardiac arrest. Prehosp Emerg Care. 2010 Oct-Dec;14(4):413-8. doi: 10.3109/10903127.2010.497902. PMID 20809686
- [Background] Salcido DD, Sundermann ML, Koller AC, Menegazzi JJ. Incidence and outcomes of rearrest following out-of-hospital cardiac arrest. Resuscitation. 2015 Jan;86:19-24. doi: 10.1016/j.resuscitation.2014.10.011. Epub 2014 Oct 23. PMID 25447433
- [Background] Jollis JG, Al-Khalidi HR, Roettig ML, Berger PB, Corbett CC, Doerfler SM, Fordyce CB, Henry TD, Hollowell L, Magdon-Ismail Z, Kochar A, McCarthy JJ, Monk L, O'Brien P, Rea TD, Shavadia J, Tamis-Holland J, Wilson BH, Ziada KM, Granger CB. Impact of Regionalization of ST-Segment-Elevation Myocardial Infarction Care on Treatment Times and Outcomes for Emergency Medical Services-Transported Patients Presenting to Hospitals With Percutaneous Coronary Intervention: Mission: Lifeline Accelerator-2. Circulation. 2018 Jan 23;137(4):376-387. doi: 10.1161/CIRCULATIONAHA.117.032446. Epub 2017 Nov 14. PMID 29138292
- [Background] Adeoye O, Nystrom KV, Yavagal DR, Luciano J, Nogueira RG, Zorowitz RD, Khalessi AA, Bushnell C, Barsan WG, Panagos P, Alberts MJ, Tiner AC, Schwamm LH, Jauch EC. Recommendations for the Establishment of Stroke Systems of Care: A 2019 Update. Stroke. 2019 Jul;50(7):e187-e210. doi: 10.1161/STR.0000000000000173. Epub 2019 May 20. PMID 31104615
- [Background] Committee on the Treatment of Cardiac Arrest: Current Status and Future Directions; Board on Health Sciences Policy; Institute of Medicine; Graham R, McCoy MA, Schultz AM, editors. Strategies to Improve Cardiac Arrest Survival: A Time to Act. Washington (DC): National Academies Press (US); 2015 Sep 29. Available from http://www.ncbi.nlm.nih.gov/books/NBK305685/ PMID 26225413
- [Background] McCarthy JJ, Carr B, Sasson C, Bobrow BJ, Callaway CW, Neumar RW, Ferrer JME, Garvey JL, Ornato JP, Gonzales L, Granger CB, Kleinman ME, Bjerke C, Nichol G; American Heart Association Emergency Cardiovascular Care Committee; Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; and the Mission: Lifeline Resuscitation Subcommittee. Out-of-Hospital Cardiac Arrest Resuscitation Systems of Care: A Scientific Statement From the American Heart Association. Circulation. 2018 May 22;137(21):e645-e660. doi: 10.1161/CIR.0000000000000557. Epub 2018 Feb 26. PMID 29483084
- [Background] Patterson T, Perkins GD, Joseph J, Wilson K, Van Dyck L, Robertson S, Nguyen H, McConkey H, Whitbread M, Fothergill R, Nevett J, Dalby M, Rakhit R, MacCarthy P, Perera D, Nolan JP, Redwood SR. A Randomised tRial of Expedited transfer to a cardiac arrest centre for non-ST elevation ventricular fibrillation out-of-hospital cardiac arrest: The ARREST pilot randomised trial. Resuscitation. 2017 Jun;115:185-191. doi: 10.1016/j.resuscitation.2017.01.020. Epub 2017 Feb 4. PMID 28174052
- [Background] Elmer J, Rittenberger JC, Coppler PJ, Guyette FX, Doshi AA, Callaway CW; Pittsburgh Post-Cardiac Arrest Service. Long-term survival benefit from treatment at a specialty center after cardiac arrest. Resuscitation. 2016 Nov;108:48-53. doi: 10.1016/j.resuscitation.2016.09.008. Epub 2016 Sep 17. PMID 27650862
- [Background] Berg KM, Cheng A, Panchal AR, Topjian AA, Aziz K, Bhanji F, Bigham BL, Hirsch KG, Hoover AV, Kurz MC, Levy A, Lin Y, Magid DJ, Mahgoub M, Peberdy MA, Rodriguez AJ, Sasson C, Lavonas EJ; Adult Basic and Advanced Life Support, Pediatric Basic and Advanced Life Support, Neonatal Life Support, and Resuscitation Education Science Writing Groups. Part 7: Systems of Care: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S580-S604. doi: 10.1161/CIR.0000000000000899. Epub 2020 Oct 21. PMID 33081524
- [Background] Anderson ML, Nichol G, Dai D, Chan PS, Thomas L, Al-Khatib SM, Berg RA, Bradley SM, Peterson ED; American Heart Association's Get With the Guidelines-Resuscitation Investigators. Association Between Hospital Process Composite Performance and Patient Outcomes After In-Hospital Cardiac Arrest Care. JAMA Cardiol. 2016 Apr 1;1(1):37-45. doi: 10.1001/jamacardio.2015.0275. PMID 27437652
- [Background] Stub D, Schmicker RH, Anderson ML, Callaway CW, Daya MR, Sayre MR, Elmer J, Grunau BE, Aufderheide TP, Lin S, Buick JE, Zive D, Peterson ED, Nichol G; ROC Investigators. Association between hospital post-resuscitative performance and clinical outcomes after out-of-hospital cardiac arrest. Resuscitation. 2015 Jul;92:45-52. doi: 10.1016/j.resuscitation.2015.04.015. Epub 2015 Apr 24. PMID 25917263
- [Background] Kurz MC, Donnelly JP, Wang HE. Variations in survival after cardiac arrest among academic medical center-affiliated hospitals. PLoS One. 2017 Jun 5;12(6):e0178793. doi: 10.1371/journal.pone.0178793. eCollection 2017. PMID 28582400
- [Background] Huebinger R, Thomas J, Abella BS, Waller-Delarosa J, Al-Araji R, Witkov R, Villa N, Nikonowicz P, Renbarger T, Panczyk M, Bobrow B. Impact of post-arrest care variation on hospital performance after out-of-hospital cardiac arrest. Resusc Plus. 2022 Apr 5;10:100231. doi: 10.1016/j.resplu.2022.100231. eCollection 2022 Jun. PMID 35434670
- [Background] Coute RA, Nathanson BH, Mader TJ, McNally B, Kurz MC. Trend analysis of disability-adjusted life years following adult out-of-hospital cardiac arrest in the United States: A study from the CARES Surveillance Group. Resuscitation. 2021 Jun;163:124-129. doi: 10.1016/j.resuscitation.2020.10.048. Epub 2020 Dec 29. PMID 33359108
- [Background] Coute RA, Nathanson BH, Kurz MC, DeMasi S, McNally B, Mader TJ. Annual and lifetime economic productivity loss due to adult out-of-hospital cardiac arrest in the United States: A study for the CARES Surveillance Group. Resuscitation. 2021 Oct;167:111-117. doi: 10.1016/j.resuscitation.2021.07.034. Epub 2021 Aug 10. PMID 34389450
- [Background] Gowens P, Smith K, Clegg G, Williams B, Nehme Z. Global variation in the incidence and outcome of emergency medical services witnessed out-of-hospital cardiac arrest: A systematic review and meta-analysis. Resuscitation. 2022 Jun;175:120-132. doi: 10.1016/j.resuscitation.2022.03.026. Epub 2022 Mar 30. PMID 35367317
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Anderson CAM, Arora P, Avery CL, Baker-Smith CM, Beaton AZ, Boehme AK, Buxton AE, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Fugar S, Generoso G, Heard DG, Hiremath S, Ho JE, Kalani R, Kazi DS, Ko D, Levine DA, Liu J, Ma J, Magnani JW, Michos ED, Mussolino ME, Navaneethan SD, Parikh NI, Poudel R, Rezk-Hanna M, Roth GA, Shah NS, St-Onge MP, Thacker EL, Virani SS, Voeks JH, Wang NY, Wong ND, Wong SS, Yaffe K, Martin SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2023 Update: A Report From the American Heart Association. Circulation. 2023 Feb 21;147(8):e93-e621. doi: 10.1161/CIR.0000000000001123. Epub 2023 Jan 25. PMID 36695182
- See also: Resuscitation Standards for Hospitals - R3 Report. The Joint Commission, 2022. (Accessed Nov 10, 2022 — https://www.jointcommission.org/standards/r3-report/r3-report-issue-29-resuscitation-standards-for-hospitals/